CLINICAL TRIAL: NCT00149487
Title: Randomized Controlled Trial of Problem Solving Intervention to Enhance Treatment Adherence in Pediatric Asthma
Brief Title: Enhancing Treatment Adherence in Pediatric Asthma With a Problem Solving Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 257; R01HL069547 (NIH)
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2022-09-19 (Actual); Status verified 2006-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Examination of the efficacy of a tailored problem-solving intervention compared with family-based education in improving adherence to treatment regimens for children diagnosed as having asthma and their caregivers
Who Masked: Investigator

ARMS (2):
- Experimental: Tailored Problem Solving Intervention (Experimental): Participants will be randomized to follow a tailored problem solving intervention for the child.
  Interventions: Behavioral: Tailored Problem Solving Intervention; Behavioral: Family Education Intervention
- Control: Family Education Intervention (Active Comparator): Participants will be randomized to follow a family education intervention.
  Interventions: Behavioral: Tailored Problem Solving Intervention; Behavioral: Family Education Intervention

INTERVENTIONS:
Behavioral: Tailored Problem Solving Intervention
Behavioral: Family Education Intervention

SUMMARY:
The purpose of this study is to determine the effectiveness of a tailored problem solving intervention in increasing adherence to asthma management behaviors in African American adolescents with asthma.

DETAILED DESCRIPTION:
BACKGROUND:

Children and adolescents who are unable to adhere to their medical regimen for the management of chronic illness present considerable challenges to health care providers and researchers. Pediatric asthma is a chronic illness where the consequences of non-adherence are particularly detrimental and widespread, especially among economically disadvantaged minority children and their families. Studies of intervention of asthma management are needed for this population.

DESIGN NARRATIVE:

The aim of the proposed study is to test the efficacy of a problem solving intervention that is tailored to the observed adherence behaviors and identified barriers to increasing adherence in African American children and adolescents with asthma, and their families. Patients are randomized to either a Tailored Problem Solving Intervention, or a control group who will receive Family Education Intervention. Duration of the intervention is four months.

ELIGIBILITY:
Inclusion Criteria:

* African American
* Family income to be below the poverty line
* Physician-based diagnosis of asthma of at least 12 months
* Moderate to severe asthma (moderate asthma includes daily symptoms, daily use of inhaled short acting beta-agonist, exacerbations greater than 2 times per week that affect activity, and nighttime symptoms greater than once a week, FEV1 or Peak Flow PEF between 60 and 80 percent predicted and PEF variability greater than 30 percent; severe asthma includes continual symptoms, limited physical activity, frequent exacerbations together with frequent nighttime symptoms, FEV1 or PEF less than 60 percent predicted, and PEF variability greater than 30 percent)
* Likely to be on a stable and daily medication (inhaled steroid) that can be modified electronically for the time period required to participate in the study

Exclusion Criteria:

* Presence of a serious comorbid chronic condition

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2001-01-22 (Actual); Primary Completion 2002-07-02 (Actual); Study Completion 2005-07-31 (Actual)

PRIMARY OUTCOMES:
Adherence to medical treatment, based on electronic monitors | 3, 6, 9 and 12 months
  describe the trajectories of adherence to daily inhaled corticosteroid (ICS) medication for a year in economically disadvantaged, African-American youth with asthma based on growth curve modeling

SECONDARY OUTCOMES:
Asthma-related morbidity, including symptoms, pulmonary functioning, and health-related quality of life | 3, 6, 9 and 12 months
  test the relationship of treatment adherence to symptom control, quick-relief medication, and healthcare utilization.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Drotar, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States